CLINICAL TRIAL: NCT03746236
Title: Transpulmonary Pressure Under Conditions of Increased Intra-abdominal Pressure From Pneumoperitoneum and Steep Trendelenburg
Brief Title: Transpulmonary Pressure Under Stressing Conditions
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Regina Elena Cancer Institute (Other)
Responsible Party: Principal Investigator, Ester Forastiere, Head of Department of Anaestesiology and Critical Care, Regina Elena Cancer Institute
Other Study IDs: RS1138/18
Record Dates: First submitted 2018-11-14; First posted 2018-11-19 (Actual); Last update posted 2019-09-11 (Actual); Status verified 2018-11

CONDITIONS: Ventilator-Induced Lung Injury
MeSH Terms: conditions — Ventilator-Induced Lung Injury

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Study aims to prospectively evaluate if the pressures normally applied during mechanical ventilation in laparoscopic surgery induce stress on the pulmonary wall. To do this is used measure the variation of esophageal pressure, as indirect index of the pleural pressure and therefore of the transpulmonary pressure, in response to changes in airway pressures in a group of patients undergoing robotic assisted radical prostatectomy or videolaparoscopy.

ELIGIBILITY:
Inclusion Criteria:

* ASA (american society of anesthesiologists) score ≤ III
* Patients underwent laparoscopic prostatectomy

Exclusion Criteria:

* BMI (body mass index) ≥ 30
* Impossibility to insert nasogastric tube
* Anatomic rib cage alterations

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients underwent laparoscopic or robotic assisted radical prostatectomy
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2018-11-14 (Actual); Primary Completion 2019-12-30 (Estimated); Study Completion 2019-12-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of postoperative acute complications | 24 hours
  Evaluation of pulmonary alterations using pre and postoperative ultrasonographic visualization
Dosage of inflammatory mediators | 24 hours
  Dosage of metalloproteinase and interleukin 8 in bronchoaspiration

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - Regina Elena National Cancer Institute, Rome, Rm
  - Regina Elena National Cancer Institute, Rome